CLINICAL TRIAL: NCT03143738
Title: Continuous Adductor Canal Block in Comparison to Continuous Femoral Nerve Block in Patients After Total Knee Arthroplasty: Randomized Control Trail
Brief Title: Comparison of Regional Anesthesia Techniques After Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Lublin (Other)
Collaborators: Konskie Specjalist Hospital (Unknown)
Responsible Party: Principal Investigator, Michał Borys, associate professor, Medical University of Lublin
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KE-0254/188/2016
Record Dates: First submitted 2017-05-03; First posted 2017-05-08 (Actual); Last update posted 2019-02-28 (Actual); Status verified 2019-02

CONDITIONS: Pain, Acute; Knee Arthropathy; Postoperative Pain; Mobility Limitation
Keywords: regional anesthesia; knee replacement; pain treatment; rehabilitation
MeSH Terms: conditions — Acute Pain; Pain, Postoperative; Mobility Limitation; Agnosia | interventions — Anesthesia, Spinal

STUDY DESIGN:
Intervention Model Description: Two groups of patients randomly allocated: adductor canal group or femoral nerve group
Who Masked: Participant
Masking Description: Participants not aware of the type of continuous blockade.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- continuous anesthesia of adductor canal (Experimental)
  Interventions: Procedure: continuous anesthesia of adductor canal; Procedure: Spinal anesthesia
- continuous anesthesia of femoral nerve (Experimental)
  Interventions: Procedure: continuous anesthesia of femoral nerve; Procedure: Spinal anesthesia

INTERVENTIONS:
Procedure: continuous anesthesia of adductor canal — After subarachnoid anesthesia, but before the beginning of surgery, a catheter will be implemented to the adductor canal and infusion of 5 mL/h of 0.2 % ropivacaine will be started.
  Arms: continuous anesthesia of adductor canal
Procedure: continuous anesthesia of femoral nerve — After subarachnoid anesthesia, but before the beginning of surgery, a catheter will be implemented next to the femoral nerve (below inguinal ligament) and infusion of 5 mL/h of 0.2 % ropivacaine will be started.
  Arms: continuous anesthesia of femoral nerve
Procedure: Spinal anesthesia — Before the beginning of surgery all patients will be anesthetised with 0.5 % hyperbaric bupivacaine (Marcaine Heavy), 2.0 - 2.5 mL solution. Pencil point spinal needle will be used.
  Other Names: Subarachnoid anesthesia

SUMMARY:
Comparison of continuous adductor canal block to continuous femoral nerve block in patients after total knee arthroplasty.

All patients will be anesthetized with spinal anesthesia. Continuous infusion of ropivacaine with a catheter implemented to the adductor canal or next to the femoral nerve.

The observed goals: pain intensity, the beginning and quality of rehabilitation.

DETAILED DESCRIPTION:
Written consent will be obtained a day before the surgery. Only subarachnoidally anaesthetised patients may participate in the study. Pencil-point spinal needle and bupivacaine (Marcaine Heavy Spinal 0.5 %) will be used.

Before the beginning of operation, under ultrasound control, a catheter will be implemented to one of the chosen position: the adductor canal (the middle or lower third of thigh) or near the femoral nerve (below the inguinal ligament). The local anesthetic solution of 0.2 % ropivacaine will be started with an elastomeric pump (5 mL per hour, up to 72 hours) as soon as a catheter in the right position.

The pain will be measured with VAS (visual-analogue scale) 8, 24 and 48 hours after the end of operation, and at the discharge. At the same time, i.e.: 8, 24 and 48 hours from the end of surgery, the range of flexion and extension in the operated knee will be assessed. Moreover, the possibility of patient's sitting, standing up and walking will be noted.

All parameters will be reassessed before patients' discharge from the hospital. Each patient will receive paracetamol (1.0) and metamizol (1.0) intravenously (i.v.) q6h. 5 mg of morphine may be given as required, up to 2 dosages per day as a rescue medication.

ELIGIBILITY:
Inclusion Criteria:

* knee arthroplasty
* obtained consent
* subarachnoid anaesthesia

Exclusion Criteria:

* coagulopathy
* allergy to to local anesthetics
* depression, antidepressant drugs treatment
* epilepsy
* usage of painkiller before surgery
* addiction to alcohol or recreational drugs

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-04-24 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-07-26 (Actual)

PRIMARY OUTCOMES:
Morphine consumption | 24 hours from the end of surgery
  Total consumption of intravenous morphine by patients with the use of patient-controlled analgesia pump

SECONDARY OUTCOMES:
Knee flexion | 8, 24, 48 hours from the end of surgery, and at the patient discharge from the hospital (an average 4-6 days)
  range of flexion in operated knee
Walking | 8, 24, 48 hours from the end of surgery, and at the patient discharge from the hospital (an average 4-6 days)
  Possibility of walking by patients at scheduled time points
The change of acute postoperative pain | 8, 24, 48 hours from the end of surgery, and at the patient discharge from the hospital (an average 4-6 days)
  Measured with VAS (visual-analogue scale)
Sitting | 8, 24, 48 hours from the end of surgery, and at the patient discharge from the hospital (an average 4-6 days)
  Possibility of walking by patients at scheduled time points

CONTACTS AND LOCATIONS:
Overall Officials: Michał Borys, M.D., PhD, Principal Investigator — Medical University of Lublin
Locations (1):
- Michał Borys, Lublin, Poland

IPD SHARING:
Plan to Share IPD: No